CLINICAL TRIAL: NCT03420807
Title: Evaluation of Beta-amyloid Plaques of the Retina Using Metabolic Hyperspectral Retinal Camera (MHRC) in Alzheimer's Patients - Toronto Study Arm
Brief Title: Retinal Metabolic Imaging of Alzheimer Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Optina Diagnostics Inc. (Industry)
Collaborators: McGill University (Other); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 071317
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Subjects will undergo 1) clinical characterization, 2) ophthalmic evaluation, 3) evaluation with the device (camera) and 4) brain imaging session (MRI + amyloid PET).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MHRC camera (Experimental): Subjects will undergo a retina imaging session with the MHRC camera.
  Interventions: Device: MHRC

INTERVENTIONS:
Device: MHRC — Evaluate the feasibility of detection of beta-amyloid plaques by using their spectral signature in autofluorescence or reflectance.

SUMMARY:
This research project concerns the evaluation of the Metabolic Hyperspectral Retinal Camera (MHRC), a novel medical instrument from Optina Diagnostics, for the detection of beta-amyloid plaques, a hallmark of Alzheimer's disease (AD), in the retina. The experimental device, produces multiple images of the retina when subjected to light in very specific colors (90-100 specific colors typically) and may be used to identify specific biomarkers based on their unique spectral signature. The retina is an extension of the brain and is the only optically accessible nervous tissue. The MHRC could represent a simple and non-invasive tool to facilitate the diagnosis of AD.

DETAILED DESCRIPTION:
Alzheimer's disease (AD), a neurodegenerative disorder characterized by cognitive impairment and a suspected dementia syndrome, is the most common type of dementia (>50% of all cases), affecting millions worldwide, with no cure available at this time. Definite AD diagnosis currently relies on the post-mortem observation of the hallmarks β-amyloid peptides (Aβ) extracellular aggregates, Aβ plaques, and protein tau intracellular twisted strands (neurofibrillary tangles, NFTs). Earlier diagnosis could dramatically transform the design and execution of clinical trials to test new treatments. The eye offers a natural window to the brain as the retina, the light sensitive layer lining the interior of the eye is an extension of the brain. The presence of Aβ plaques in the retina of AD mice models and humans was recently reported opening the possibility of detecting this AD hallmark though a simple non-invasive eye scan. The proposed research aims to explore this avenue with the development of a spectrally-resolved optical retinal imaging platform to detect Aβ plaques in the retina of AD subjects and validate the method against brain Aβ plaques seen on amyloid PET imaging. The novel imaging platform is expected to help aid the early detection of AD and assist in monitoring efficacy of possible future therapeutic agents that target relevant molecular pathways.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with Alzheimer's disease

   * Meet criteria for probable, possible Alzheimer's disease by McKhann criteria (McKhann et al. 2011)
   * Mini-Mental State Examination score between 20 and 27 (inclusive)
   * Vascular load scale ≤ 4 (Hachinski Ischaemia Score)
   * Sufficient degree of cooperation to undergo all examinations
   * Availability of a reliable responsible study partner to accompany the patient to the appointments
2. Subjects with Mild Cognitive Impairment

   * Meet criteria for amnestic single or multi domain Mild Cognitive Impairment (without crossing the threshold for dementia)
   * No signs of systemic, neurologic or psychiatric disorders that can cause cognitive deficits
   * Scores on cognitive tests: 1 to 1.5 standard deviation below the mean of their age and education matched peers
   * Diagnosis that follows Albert criteria (Albert et al. 2011)
3. Healthy control subjects

   * No clinical signs of dementia
   * Telephone Mini-Mental State Examination score ≥ 25 or
   * MoCA ≥ 26
   * Behavioural Neurology Assessment-R (BNA-R; Annex IX; within limits on all sub tests)

Exclusion Criteria:

* Presence of one or more contraindications (PET and/or MRI)
* Presence of glaucoma or retinopathy (diabetic, macular degeneration)
* Pupil dilation inadequate or contraindicated
* Deficient visual fixation
* Refractive error outside the range -9 to +9
* Impossibility of obtaining satisfactory, quality images with MHRC

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Retinal beta-amyloid detection | Within 21 days following clinical characterization completion
  Presence of absence of beta-amyloid plaques in the retina

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Black, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No